CLINICAL TRIAL: NCT00455247
Title: Efficacy of an Oral Formula in Prevention of Anti-cancer Therapy Side Effects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06.23.CLI
Record Dates: First submitted 2007-03-01; First posted 2007-04-03 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Digestive Cancers
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Glutamine

INTERVENTIONS:
Drug: Glutamine

SUMMARY:
Anti-cancer treatment is often inducing side-effects that can affect the compliance to the treatment protocol and quality of life of the patients. The researchers will study if the nutritional intervention with the product could abrogate the undesired effects in a preventive manner.

ELIGIBILITY:
Inclusion Criteria:

* Patient with GI neoplasm
* Patient that must start a (new) line of chemotherapy with at least 2 cycles
* Age > 18 ans
* Exclusively orally fed
* Life expectancy more than 3 months
* Intravenous 5FU-based chemotherapy with 2 or 3-week cycles
* Hematological toxicities from previous chemotherapies terminated or <= 2

Exclusion Criteria:

* Positive HIV status
* Pregnant or lactating woman
* Currently participating or having participated in another clinical trial during the last month prior to the beginning of this study
* Patient having diarrhoea of grade > 1 for more than 2 weeks before the inclusion
* State of sub occlusion, chronic inflammatory diseases of the digestive tract, radiation enteropathy
* Sepsis
* Concomitant radiotherapy, except analgesic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SENESSE, MD, Principal Investigator — CRLC Val d'Aurelle
Locations (7):
- France (7):
  - Institut Sainte-Catherine, Avignon
  - CH Béziers, Béziers
  - CRLCC Léon Bérard, Lyon
  - CRLC Val d'Aurelle, Montpellier
  - CHU Montpellier, Montpellier
  - CH Perpignan, Perpignan
  - CHU Charles Nicolle, Rouen